CLINICAL TRIAL: NCT04722679
Title: BELgian ANtiCoagulation Survey for Elderly Patients With NVAF
Brief Title: A Study to Collect Information on the Characteristics of Elderly Belgian Patients With NVAF That Are Treated With a NOAC for This Indication With a Special Focus on Their Fear of Bleeding While Using a NOAC vs the Clinical Benefit of a NOAC of Thrombosis/Stroke Prevention.
Acronym: BELANCE
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21740
Record Dates: First submitted 2021-01-21; First posted 2021-01-25 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Non-Valvular Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: Elderly (defined as the ≥75 years old) patients with NVAF that are treated with a NOAC.
  Interventions: Drug: Non-VKA Oral Anticoagulants (NOAC)
- Physician: Geriatricians (hospital or office-based).
  Interventions: Drug: Non-VKA Oral Anticoagulants (NOAC)

INTERVENTIONS:
Drug: Non-VKA Oral Anticoagulants (NOAC) — Follow clinical practice.

SUMMARY:
Atrial fibrillation is a heart condition that causes an abnormal and fast heart rate. For people with non-valvular atrial fibrillation (NVAF), this is caused by problems such as high blood pressure and diabetes. NVAF happens more often in elderly people and can lead to stroke, heart failure, and death. Doctors are currently able to give patients a type of treatment called an anticoagulant. Anticoagulants work by making the blood thinner. They are thought to help reduce the risk of stroke and death caused by NVAF. In this study, researchers wanted to learn more about what elderly people think of taking anticoagulants that do not have any vitamin K in them. These are called non-VKA oral anticoagulants (NOACs).

This study will include up to about 150 Belgian men and women aged 75 years and over who have NVAF and have been treated with NOACs. The study will also include about 10 doctors who have treated these patients.

In this study, there will be no required tests or visits. Instead, patients will answer a paper questionnaire about their use of NOACs. The researchers will ask the doctors questions about how they treat their patients using NOACs. The main types of questions the researchers will focus on are:

* The patient characteristics of the elderly with NVAF who are treated with NOACs
* The level of fear of the elderly about bleeding while using a blood thinner and the fear of stroke/thrombosis.
* The geriatrician's thoughts about using NOACs to treat NVAF in elderly patients
* Those patient characteristics geriatrician's find most important when deciding on the anticoagulation treatment in the elderly patients.

The information from this study will be collected between February and April 2021. But, the whole study will take about 6 months to finish and is expected to end in July 2021.

ELIGIBILITY:
Inclusion Criteria:

* Male or female elderly patients (defined as ≥ 75 years old) diagnosed with NVAF
* Elderly patients treated with a NOAC
* Ambulatory patients visiting the geriatrician

Exclusion Criteria:

* Contra-indications according to the local marketing authorization
* Patients suffering from dementia who are, according to the geriatrician's opinion, not able to understand and answer the questions
* Hospitalized patients

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The source population of this study would be elderly patients population (defined as ≥ 75 years old) diagnosed with NVAF who are treated with a NOAC for this indication. In order to ensure the representativeness of the study population, 100-150 Belgian elderly patients will be taken into account.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-03 (Actual)

PRIMARY OUTCOMES:
Age categories of patients and the geriatricians | Approximate 3 months for data collection
Gender of patients and the geriatricians | Approximate 3 months for data collection
Patient's weight | Approximate 3 months for data collection
Patient's kidney function range (normal, mild, moderate, severe) | Approximate 3 months for data collection
CHA₂DS₂-VASc range | Approximate 3 months for data collection
  CHA2DS2-VASc score is a clinical prediction rule for estimating the risk of stroke in patients with non-rheumatic atrial fibrillation (AF), a common and serious heart arrhythmia associated with thromboembolic stroke.
Clinical Frailty Scale (CFS) range | Approximate 3 months for data collection
Timeframe of patient's diagnosis with NVAF | Approximate 3 months for data collection
Specification of HCP that initiated the elderly patient's NOAC treatment | Approximate 3 months for data collection
  HCP: HealthCare Professionals
Specification of NOAC treatment | Approximately 3 months for data collection
Use of low-dose NOAC treatment (not related to an (S)AE) | Approximate 3 months for data collection
Confirmation of the use of anti-aggregants | Approximate 3 months for data collection
Level of agreement with various statements regarding the use of NOACs in general, using a 5-point Likert scale (completely disagree, more likely to disagree, no opinion, more likely to agree, completely agree) | Approximate 3 months for data collection
Indication of fear of contracting a bleeding while using a blood thinner on a scale from 0 - 10 | Approximate 3 months for data collection
Indication of fear of contracting a stroke or thrombosis on a scale from 0 - 10 | Approximate 3 months for data collection

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.